CLINICAL TRIAL: NCT05219903
Title: National, Multicenter, Retrospective, Prospective Study to Evaluate Pediatric Gastrointestinal Eosinophilic Disorders
Acronym: GOLDEN
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Collaborators: Italian Society of Pediatric Allergy & Immunology - Pediatric Centers (Unknown)
Responsible Party: Principal Investigator, Amelia Licari, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: GOLDEN
Record Dates: First submitted 2022-01-21; First posted 2022-02-02 (Actual); Last update posted 2024-07-25 (Actual); Status verified 2024-07

CONDITIONS: Eosinophilic Gastrointestinal Disorders; Eosinophilic Esophagitis; Eosinophilic Gastritis or Gastroenteritis; Eosinophilic Colitis
Keywords: Eosinophilic gastrointestinal disorders; Children; Prevalence; Incidence
MeSH Terms: conditions — Eosinophilic Esophagitis; Eosinophilic enteropathy; Gastroenteritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Eosinophilic gastrointestinal disorders (EGIDs) are a heterogeneous group of emerging chronic inflammatory diseases that may affect different gastrointestinal (GI) tracts. Based on the anatomical site involved, EGIDs are distinguished into eosinophilic esophagitis (EoE) and non-esophageal forms, which are subdivided into eosinophilic gastritis (EoG), gastroenteritis (EoGE), and colitis (EoC). EoE is considered the prototype of EGIDs. Since the first description of a case series of patients with EoE, fundamental scientific advances have been achieved, culminating in the redaction of international diagnostic and therapeutic guidelines. In contrast to EoE, non-esophageal forms of EGIDs are still a clinical enigma with evidence limited to a few retrospective studies. In the last decade, an increase in the prevalence of EGIDs has been observed in the pediatric age. Unfortunately, the epidemiology of EGIDs in Italy is still inconsistent and clear estimates are not available.

Firstly, this study will allow us to assess and clarify several clinical and epidemiological aspects of pediatric EGIDs, in particular:

1. prevalence and incidence of pediatric EGIDs in Italy,
2. the clinical features and potential phenotypes of pediatric EGIDs with potential impact on therapy and management,
3. diagnostic work-up and adherence to the EoE international guidelines to improve the management, quality of care, and quality of life of affected patients.

This study has no ethical problems since EoE patients are treated according to international guidelines and those with non-esophageal EGIDs according to the latest scientific evidence.

ELIGIBILITY:
Inclusion Criteria:

- All EGIDs patients aged 0-18 years and followed at the centers involved in the study will be considered eligible. Informed consent must be obtained from each enrolled patient and signed by a parent/legal guardian and patient (when older than six years).

Exclusion Criteria:

- This study will not include patients with:

1. a diagnosis of EGIDs made more than five years before the study participation;
2. a diagnosis of EoE not in line with current international guidelines;
3. a secondary cause of intestinal eosinophilic inflammation (inflammatory bowel diseases, autoimmune diseases, vasculitis, graft versus host disease, malignancies).

Ages: 0 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: EoE and EGIDs Definition: Based on current international guidelines, EoE diagnosis requires the presence of more than 15 eos/HPF in endoscopically obtained esophageal biopsies.5 In contrast, the diagnosis of non-esophageal EGIDs should meet the following criteria:
  * Chronic/recurrent GI symptoms unresponsive to standard therapies,
  * A prevalent eosinophilic intestinal inflammation,
  * Exclusion of secondary causes of intestinal eosinophilia (e.g., intestinal parasitosis, chronic inflammatory bowel disease, vasculitis, autoimmune diseases, graft versus host disease, tumors).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence estimates | 5 years
  a) To estimate the EGIDs prevalence in patients with gastrointestinal symptoms undergoing upper and lower GI endoscopy, to verify whether the global increase of EGIDs also affects the Italian reality
Incidence estimates | 5 years
  b) If available the cumulative incidence (new EGIDs cases) may be derived, as a subgroup analysis of the primary endpoint
Prospective epidemiological estimates | 5 years
  a) To estimate the cumulative incidence of EGIDs (new diagnosis of EGIDs) over the study period.

SECONDARY OUTCOMES:
Other epidemiological estimates | 5 years
  a) To compare the cumulative incidence of EGIDs observed in the prospective with the data from the retrospective study (if available) and those available in the literature, to verify the increase of EGIDs, previously observed in a few US observational studies;
Definition of clinical features and potential phenotypes | 5 years
  b) To describe the clinical characteristics of Italian patients with EGIDs (risk factors, sex, age, comorbidities, response to therapy, natural history), to identify potential phenotypes;
Improvement of diagnostic and therapeutic management | 5 years
  c) To define shared diagnostic-therapeutic management and verify the adherence of enrolled centers to the international EoE guidelines.

CONTACTS AND LOCATIONS:
Overall Officials: Amelia Licari, MD, Study Director — IRCCS Policlinico San Matteo
Locations (1):
- IRCCS Policlinico San Matteo, Pavia, Italy

REFERENCES:
- [Background] Licari A, Votto M, Scudeller L, De Silvestri A, Rebuffi C, Cianferoni A, Marseglia GL. Epidemiology of Nonesophageal Eosinophilic Gastrointestinal Diseases in Symptomatic Patients: A Systematic Review and Meta-Analysis. J Allergy Clin Immunol Pract. 2020 Jun;8(6):1994-2003.e2. doi: 10.1016/j.jaip.2020.01.060. Epub 2020 Feb 28. PMID 32061717
- [Background] Licari A, Votto M, D'Auria E, Castagnoli R, Caimmi SME, Marseglia GL. Eosinophilic Gastrointestinal Diseases in Children: A Practical Review. Curr Pediatr Rev. 2020;16(2):106-114. doi: 10.2174/1573396315666191022154432. PMID 31642786
- [Background] Votto M, Castagnoli R, De Filippo M, Brambilla I, Cuppari C, Marseglia GL, Licari A. Behavioral issues and quality of life in children with eosinophilic esophagitis. Minerva Pediatr. 2020 Oct;72(5):424-432. doi: 10.23736/S0026-4946.20.05913-7. Epub 2020 Jun 4. PMID 32506880
- [Background] Votto M, Marseglia GL, De Filippo M, Brambilla I, Caimmi SME, Licari A. Early Life Risk Factors in Pediatric EoE: Could We Prevent This Modern Disease? Front Pediatr. 2020 May 29;8:263. doi: 10.3389/fped.2020.00263. eCollection 2020. PMID 32548083
- [Background] Votto M, De Filippo M, Olivero F, Raffaele A, Cereda E, De Amici M, Testa G, Marseglia GL, Licari A. Malnutrition in Eosinophilic Gastrointestinal Disorders. Nutrients. 2020 Dec 31;13(1):128. doi: 10.3390/nu13010128. PMID 33396413
- [Background] Votto M, Raffaele A, De Filippo M, Caimmi S, Brunero M, Riccipetitoni G, Marseglia GL, Licari A. Eosinophilic gastrointestinal disorders in children and adolescents: A single-center experience. Dig Liver Dis. 2022 Feb;54(2):214-220. doi: 10.1016/j.dld.2021.06.027. Epub 2021 Jul 15. PMID 34274254